CLINICAL TRIAL: NCT06870344
Title: After the Flood: Optimal Strategies to Prevent Malaria Epidemics Caused by Severe Flooding
Brief Title: IGHID 12334 - After the Flood: Optimal Strategies to Prevent Malaria Epidemics Caused by Severe Flooding
Acronym: IGHID12334
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); North Carolina State University (Other); Mbarara University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24-0233; 1R01AI173558-01A1 (NIH)
Record Dates: First submitted 2025-03-03; First posted 2025-03-11 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Malaria Infection; Malaria Falciparum
Keywords: Flooding, malaria incidence; malaria; plasmodium
MeSH Terms: conditions — Malaria, Falciparum; Malaria

STUDY DESIGN:
Intervention Model Description: The study is an open-label, cluster randomized controlled trial. randomized 1:1:1 within each stratum to either control (i.e., LLIN only) or one of the two intervention groups (DP or DP+Bti).
  Control - LLIN distribution Arm 1 - LLIN + monthly DP for children ≤12 years of age Arm 2 - LLIN + DP + Bti
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Arm: Provision of new Long-lasting Insecticidal Net (LLIN(s) the participant household (Other): Control Arm: Provision of new LLIN(s) to bring the household up to WHO "universal coverage" targets defined as one LLIN per every two household residents.
  Interventions: Other: Long-lasting Insecticidal Net
- Dihydroartemisinin Piperaquine (DP) (Active Comparator): LLIN + monthly DP for children ≤12 years of age In addition to receipt of LLIN(s) as described above, children ≥2 to ≤12 years of age will be screened for DP administration. If no contraindications are noted, weight-based DP will be administered by the parent/caregiver under the supervision of the study team. Participants will be observed for ~ 30 minutes. Any adverse events will be documented. Tablets for administration on Days 2 and 3 will be provided. Administration will be repeated at months 2 and 3 post-flooding.
  Interventions: Drug: Dihydroartemisinin piperaquine
- Dihydroartemisinin Piperaquine(DP)+Bacillus thuringiensis israelensis(Bti) (Active Comparator): LLIN + DP + Bti In addition to receipt of LLIN(s) and DP, study staff will provide the adult participant with an 8-oz packet of Bti, a pair of latex gloves, a teaspoon, and a tracking form. A staff member will then survey an area (50 m radius) around the house and demonstrate appropriate application in up to 5 potential breeding sites. Household members will be instructed to repeat application every 2 weeks for the 3 months post-flooding.
  Interventions: Combination Product: Dihydroartemisinin piperaquine + Bacillus thuringiensis israelensis

INTERVENTIONS:
Drug: Dihydroartemisinin piperaquine — Taken orally. 11 kg to less than 17 kg 1 tablet per day for 3 days 40 mg 320 mg 17 kg to less than 25 kg 1½ tablets per day for 3 days 60 mg 480 mg 25 kg to less than 36 kg 2 tablets per day for 3 days 80 mg 640 mg 36 kg to less than 60 kg 3 tablets per day for 3 days 120 mg 960 mg 60 kg to less than 80 kg 4 tablets per day for 3 days 160 mg 1280 mg 80 kg or more 5 tablets per day for 3 days 200 mg 1600 mg For patients weighing less than 11 kg, alternative formulations supplying lower amounts of active substance should be preferred
  Other Names: Eurartesim
  Arms: Dihydroartemisinin Piperaquine (DP)
Combination Product: Dihydroartemisinin piperaquine + Bacillus thuringiensis israelensis — Study staff will provide adult participant with LLIN(s), DP and with an 8-oz packet of Bti, a pair of latex gloves, a teaspoon, and a tracking form. A staff member will then survey an area (50 m radius) around the house and demonstrate appropriate application in up to 5 potential breeding sites.
  Arms: Dihydroartemisinin Piperaquine(DP)+Bacillus thuringiensis israelensis(Bti)
Other: Long-lasting Insecticidal Net — Distribution of Long-lasting Insecticidal Net to all households on the study.
  Other Names: bed nets
  Arms: Control Arm: Provision of new Long-lasting Insecticidal Net (LLIN(s) the participant household

SUMMARY:
The purpose of this study is to test different ways to prevent malaria infections after flooding. To accomplish this, the investigators will assign villages to different control strategies and measure the number of malaria infections in each of the villages. Residents of all villages will receive new bed nets, but in some villages, residents will be provided with a monthly medication Dihydroartemisinin-piperaquine (DP) (a drug that is approved by the World Health Organization (WHO) and regulatory authorities and widely used in Africa for Malaria treatment. This drug is not approved by Food and Drug Administration (FDA) because it is not used in the US,) to prevent malaria, while others will also receive a treatment that can be placed into pools of water around the home to prevent mosquitoes from breeding there. The investigators will monitor the participant and their household members for mosquitoes and malaria over a period of 12 months after the flooding This study is important because, similar approaches could be used to prevent malaria after floods, which is occurring more frequently.

DETAILED DESCRIPTION:
The study is an open-label, cluster randomized controlled trial in fifty villages prone to predictable, but often catastrophic annual flooding in a malaria-endemic area of western Uganda.

STUDY DESIGN The investigators will conduct an open-label, cluster randomized controlled trial in approximately 50-60 villages prone to predictable, but often catastrophic annual flooding in a malaria-endemic area of western Uganda. In the first year, the investigators will conduct baseline surveys of participating households, including geographic variables (e.g., elevation, proximity to river) and measures such as malaria transmission intensity (Plasmodium falciparum Positivity Rate (PfPR)) to stratify risk. The unit of randomization will be the sub-village, defined as the geographic area of responsibility for each community health worker, typically comprised of approximately 200-300 residents living in 30-40 distinct households. The N=144 sub-village (clusters) will be stratified based on pre-flood malaria transmission intensity and randomized 1:1:1 within each stratum to either control (i.e.,Long-lasting Insecticidal Net (LLIN only)) or one of the two intervention groups (DP or DP+Bti). Participants will be followed longitudinally for a period of 12-months after the index flood event. The investigators will conduct facility-based surveillance for parasitologically-confirmed, symptomatic malaria cases, measure PfPR, assess entomological risk, and socioeconomic impacts of the intervention(s).

STUDY ENROLLMENT AND WITHDRAWAL Strategies for Recruitment and Retention Sensitization Meetings & Community Dissemination The investigators will conduct a series of sensitization meetings with sub-county and village leadership in each of the study areas to inform them of the aims and methods of the study. These meetings will be followed similar events with community health workers (CHWs), who will be asked to disseminate the information, as well as the proposed dates of the baseline surveys, to households in their respective coverage areas.

Enrollment On the day of the baseline survey, study staff, guided by the local CHW, will approach each household in the sub-village. If an adult (age ≥18 years) household member is present, study staff, fluent in Lukhonzo, will review the aims and methods of the study and ask for written consent to participate. Children 8 - 17 years of age will be asked to provide written assent. Households without an adult present will be revisited two additional times, after which the household will be geolocated, but considered not participating.

Participant Incentives

Participants will be eligible to receive the following incentives for participation:

Event Eligibility Amount (UGX) Initial Visit Visit Completed 20,000 Follow-up Visit (4) Visit Completed 5,000 Final Visit Visit Completed 10,000 POTENTIAL TOTAL 50,000

*Approximate UGX to United State Dollar (USD) conversion; may change based on exchange rate

Participating children undergoing any examination, blood draw, or medication administration will also receive an in-kind incentive such as a juice, biscuit, or similar item.

Contacts On enrollment, participants will be asked to provide the best contact information, including a mobile phone number, if available. Study staff will confirm if this phone is owned/used by the participant or belongs to someone else (e.g., neighbor, relative). In addition, the investigators will ask for permission to send reminders for upcoming study visits via text or phone call. If a participant confirms attendance, then no further contact will be made. Study staff will make up to three text or phone contacts prior to a scheduled study visit. If study staff are unable to locate participant after three attempts, staff will contact the CHW responsible for the area and request assistance contacting the participant, which may include up to three visits to the home.

Treatment Assignment Procedures Triggering Event

Due to the lack of weather monitoring equipment in the region, it is difficult to define objectively a flood event based on measures such as rainfall, river depth, or river flow. Instead, when the investigators receive reports of flooding from local communities, the nature of the flood will be investigated (i.e., rainfall, mud slide, human-caused) and extent of the flooding. Key indicators suggestive of a flood event include:

* Water overflowing established banks of the respective river
* Displacement of residents from their homes due to flooding
* Closure or damage to key infrastructure (e.g., roads, bridges, clinics) due to flooding

When an event is reported, study leadership will convene and determine if these key indicators are met, after which time a decision will be made to initiate the intervention or not. Because the extent of flooding may be limited to one river, the decision to initiate study activities may only involve sub-villages located in basin.

Randomization Procedures The trial will be conducted in 50-60 villages located along the banks of the Mubuku, Nyamwamba, and Nyamughasane Rivers in the Kasese District of western Uganda. Each village is divided into five sub-villages, defined by each CHW's area of responsibility, which will serve as the unit of randomization. Sub-villages are typically comprised of approximately 200-300 residents living in 30-40 distinct households. Sub-villages that cannot be reached by motorized transportation (e.g., motorcycle) or have minimal malaria at baseline (PfPR<5%) will be excluded. From the 250-300 possible sub-villages, the investigators will purposively select 144 sub-villages for inclusion in the study such that the number of contiguous clusters is minimized and to include sub-villages with the most severe flooding. This will be done to reduce the potential for spillover effects (i.e., the chance that an intervention administered in one sub-village will affect the rate of malaria in an adjacent sub-village). As much as possible, the research team will attempt to ensure ≥1 km between the location of each sub-village, defined as the location of the respective community health worker's household. This distance was chosen as it represents the upper range of Anopheles mosquito flight.

The N=144 clusters will be stratified based on pre-flood (baseline PfPR levels) malaria transmission intensity and river valley membership (e.g., Mubuku, Nyamwamba, or Nyamughasane) to maximize balance in flooding intensity across treatment arms. Within each stratum, clusters will be randomized in a 1:1:1 ratio between Control, DP, and DP+Bti arms. The investigators will utilize block randomization to ensure an even distribution of clusters across treatment arms within each stratum. The randomization protocol will be developed and implemented by a University of North Carolina (UNC) biostatistician not involved in the direct enrollment of participants. Participants and study staff will be aware of the allocation.

Subject Withdrawal Participants will be followed until participant closeout, withdrawal of consent, or death. A participant may withdraw from the study at any time at his/her own request or may be withdrawn at any time at the discretion of the investigator for safety, behavioral, compliance, or administrative reasons. This is expected to be uncommon. If the participant withdraws consent for disclosure of future information, the sponsor may retain and continue to use any data collected before such a withdrawal of consent.

Reasons for Withdrawal

Subjects are free to withdraw from participation in the study at any time upon request. An investigator may terminate a study subject's participation in the study if:

* Any clinical Adverse Event (AE), laboratory abnormality, or other medical condition or situation occurs such that continued participation in the study would not be in the best interest of the subject.
* The subject meets an exclusion criterion (either newly developed or not previously recognized) that precludes further study participation. This may include change of residence outside the study area.
* The subject is "lost to follow-up" defined as failure to attend three consecutive study visits and staff are unable to contact by phone or proxy.

Handling of Subject Withdrawals or Subject Discontinuation of Study Intervention Given the established safety profile of the proposed interventions there is minimal risk associated with use outside the parameters of the study. Therefore, subjects who withdraw or otherwise discontinue participation will not be followed further.

Premature Termination or Suspension of Study This study may be suspended or prematurely terminated if there is sufficient reasonable cause. Written notification, documenting the reason for study suspension or termination, will be provided by the suspending or terminating party to the sponsor and relevant regulatory authorities. If the study is prematurely terminated or suspended, the principal investigator (PI) will promptly inform the relevant IRB(s) and will provide the reason(s) for the termination or suspension.

Circumstances that may warrant termination include, but are not limited to:

* Determination of unexpected, significant, or unacceptable risk to subjects.
* Insufficient adherence to protocol requirements.
* Data that are not sufficiently complete and/or evaluable.

STUDY INTERVENTION Study Product Description Dihydroartemisinin-piperaquine (DP) is a WHO pre-qualified artemisinin combination therapy widely used for the treatment of uncomplicated malaria. Dosing is weight-based with tablets administered once a day for three days. Because of its relatively long half-life, estimated to be ~21 days, DP has also been employed for a range of chemoprevention strategies including intermittent preventative treatment programs, mass drug administration, and seasonal malaria chemoprevention. In the pilot study that provides the rationale for this trial, the investigators found that DP was both effective and well-tolerated. While the investigators do not propose administration to women of child-bearing age, DP has been demonstrated to be safe when used for the prevention of malaria in pregnancy.

The biologic larvicide Bacillus thuringiensis israelensis (Bti) is non-toxic to mammals, birds, and fish. Cases of irritation resulting from direct eye or skin exposure to Bti have been reported.

Acquisition DP will be obtained via the Joint Medical Stores (JMS), who will ensure integrity of the product. All medication will have a sufficiently long expiry (≥2 years) such that the investigators can ensure administration prior to expiration. The supply of Bti will be obtained directly from Summit Chemical (Baltimore, USA), who manufactures Mosquito Bits ® a US Environmental Protection Agency registered larvicide available in a convenient corn-sized granule.

Formulation, Packaging, and Labeling DP will be provided by the manufacturer in blister packs. Two dose packs are available, either 20/160 mg tablets or 40/320 mg tablets.

Bti granules will be provided in individual, resealable plastic bags (8 oz) in accordance with the manufacturer's standard packaging.

Product Storage and Stability In accordance with the manufacturer's instructions, DP will be stored in the original containers protected from light and moisture, not above 25 degrees celsius. All products will be used prior to expiry.

Staff and participants will be instructed to store Bti in the original container with original label in a cool, well-ventilated place away from children. In addition, the container should be closed when not in use. This material is not regulated by the U.S. Department of Transportation as a hazardous material.

ELIGIBILITY:
Inclusion Criteria:

* Permanent resident of flood-prone village in Kasese District with no plans to change residency in subsequent 12 months
* Able and willing to comply with all study procedures and be available for the duration of the study
* Able and willing to consent to study procedures as documented on informed consent form (ICF). For children (age <18 years), parent or guardian must provide consent. Children age ≥8 to 17 years will also be asked to provide written assent.

Exclusion Criteria:

* Temporary or part-time residence in study village
* Plans to move in the next 12 months
* Unable or unwilling to provide consent.
* Anything that would place the individual at increased risk or preclude the individual's full compliance with or completion of the study.

Ages: 0 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 36000 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
A. Cluster-level Incidence of malaria in children ≤ 12 years of age | up to 12 months after the flooding
  The cluster-level incidence of confirmed, symptomatic malaria in children ≤ 12 years of age, defined as fever (Temp ≥38 degrees Celsius (°C)) or a subjective history or fever in the prior 24 hours as the cause of care seeking and a positive malaria diagnostic test (i.e., Rapid Diagnostic Test (RDT) or microscopy), per 1,000 residents over the twelve-month period of observation. Incident cases will be captured at neighboring health facilities. In addition, the investigators will conduct a series of household surveys at baseline and 1-, 3-, 6-, and 12-months post-flooding in order to monitor temporal changes in the spatial distribution of malaria parasitemia, vector populations, and resulting social/economic impacts.

SECONDARY OUTCOMES:
A. Cluster-level Incidence of malaria among all residents | 1-, 3-, 6-, and 12-months post flooding.
  Acute febrile illness as previously defined AND positive RDT/microscopy at catchment health facility among all residents will be collected.
Change in prevalence of anemia in children <5 years of age | baseline, 6-, and 12 months after the flooding
  Hemoglobin concentration ≤7.0 g/dL measured in children <5 years of age using Hemocue device.
Change in WHO Indicators of Acute Malnutrition in children <5 years of age | baseline, 6, and 12-months post flooding.
  Acute malnutrition will be assessed via mid-upper arm circumference (MUAC).
Change in WHO Indicators of Chronic Malnutrition in children <5 years of age | baseline, 6, and 12-months post flooding.
  The WHO uses 3 indicators of chronic malnutrition (stunting, wasting, and underweight). This will be assessed in children <5 years as defined by any one of the following:
  * stunting - height-for-age <-2 SD of the WHO Child growth standards median;
  * wasting - weight-for-height <-2 SD of the WHO Child growth standards median; and
  * underweight - weight-for-age <-2 standard deviations (SD) of the WHO Child growth standards median
Prevalence of parasitemia in children | 1-, 3-, 6-, and 12-months post flooding.
  >RDT performed in all children ≤12 years during household surveys.
Hospitalization for malaria | 12 months after the flooding
  Self-reported history of hospitalization on bi-weekly questionnaire AND confirmation by study staff from hospital registers
Cluster-level change in Anopheles density and species composition | 12 months after the flooding
  Longitudinal surveillance of indoor and outdoor (i.e., peri-domestic) adult mosquitoes using Centers for Disease Control and Prevention (CDC) light traps
Prevalence of juvenile Anopheles within peri-domestic space | 12 months after the flooding
  Longitudinal surveys of 50 m radius around household with inspection of potential breeding sites
Cluster-level change in blood-fed and parasite-carrying Anopheles | 12 months after the flooding
  Polymerase Chain Reaction (PCR) of mosquitoes to estimate proportion with human blood and P. falciparum (i.e., sporozoite rate)
Cost-effectiveness of interventions (DP, DP+Bti) compared to control (LLINs) | 12 months after the flooding
  Incremental Disability Adjusted Life Year (DALY) averted.
Adherence to intervention components (LLIN, DP, and Bti) | 12 months after the flooding
  Self-reported bed net use the night prior to data collection; number of doses of DP administered per month over 3 month period; number of Bti applications over study period

CONTACTS AND LOCATIONS:
Overall Officials: Ross Boyce, MD, M.Sc., Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Mbarara University of Science and Technology (MUST), Mbarara, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Time Frame: beginning 9 and continuing through 36 months following publication
Access Criteria: Requesting investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.